CLINICAL TRIAL: NCT00206401
Title: Conventional Insulin Therapy Vs Intensive Insulin Management In Children With Type 1 Diabetes Mellitus
Brief Title: Lantus in the Treatment of Type 1 Diabetes Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sponsored Programs, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16559
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: Adolescents; Lantus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Lantus and short acting analogs Vs NPH and short acting analogs

SUMMARY:
In this study, we plan to examine the difference in effect on blood glucose control in patients who will be on either conventional insulin therapy (i.e. using NPH and Humalog twice daily, injected separately) or on intensive insulin management (IIM-several shots of short acting and Glargine insulin). Those on IIM will be mixing the insulin Glargine with the short-acting insulin analog prior to injecting. The Hemoglobin A1c (HbA1c) results will be used to monitor blood glucose control over a 6 month period. Twice during the course of the study, a continuous glucose monitoring system (CGMS-a device the size of a pager that records blood sugar readings every 5 minutes) will be used to record all the changes in the blood glucose levels occurring over a 72-hour period.

DETAILED DESCRIPTION:
The landmark report of the diabetes control and complications trial (DCCT) trial has shown that intensive management delays and/or prevents complications in small vessels associated with Type 1 diabetes (T1DM). To achieve the goals of the DCCT, a number of new insulin analogs( man-made insulins ) are now being incorporated into the management of patients with T1DM.

These insulin analogs are gaining importance with their ability to overcome the major obstacle to intensive insulin therapy, namely low blood glucose. In particular, insulin Glargine, considered a basal insulin, is being extensively used for management as an alternative to continuous insulin therapy injected into the tissue just below the skin. The major drawback to using insulin Glargine is that it has to be given as a separate injection and cannot be mixed with other insulins. This results in the undesirable administration of multiple insulin injections to a child with diabetes making the therapeutic plan more complex and adhering to the treatment plan more difficult.

In a previous study, (now accepted for publication in a leading diabetes journal, Diabetes Care), we have demonstrated, using continuous glucose monitoring system, that there is no significant difference in glucose concentrations (ie. high and low blood glucose episodes) when insulin Glargine is administered either mixed with a short-acting insulin analog or when giving it as a separate injection.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 6 years of age but less than 25 years of age (Insulin glargine has been approved for use in children 6 years and older).
* Patients newly diagnosed with T1DM within the past 3 months.
* Have an HgbA1c of less than 9.0%, after the initial run-in period of 3 months.
* Have a BMI of less than the 90th percentile for age.
* Randomization of subjects willing to participate in the study.

Exclusion Criteria:

* Any chronic disease (leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis, etc) that directly, or as a result of treatment, directly or indirectly affect glucose homeostasis.
* Lack of supportive family.
* Evidence or history of chemical abuse.
* Age less than 6 years or greater than 25 years.
* HbA1c level of greater than 9.0%, after the initial run-in period of 3 months.
* Have a BMI greater than the 90th percentile for age.
* Patients who are not newly diagnosed with T1DM.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2004-11; Study Completion 2006-10

PRIMARY OUTCOMES:
HbA1C

SECONDARY OUTCOMES:
Glucose excursions

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Kaplan W, Rodriguez LM, Smith OE, Haymond MW, Heptulla RA. Effects of mixing glargine and short-acting insulin analogs on glucose control. Diabetes Care. 2004 Nov;27(11):2739-40. doi: 10.2337/diacare.27.11.2739. No abstract available. PMID 15505016
- [Derived] Hassan K, Rodriguez LM, Johnson SE, Tadlock S, Heptulla RA. A randomized, controlled trial comparing twice-a-day insulin glargine mixed with rapid-acting insulin analogs versus standard neutral protamine Hagedorn (NPH) therapy in newly diagnosed type 1 diabetes. Pediatrics. 2008 Mar;121(3):e466-72. doi: 10.1542/peds.2007-1679. Epub 2008 Feb 25. PMID 18299307